CLINICAL TRIAL: NCT06037850
Title: Clinical Trial of Orthokeratology Lens (MCOK-01)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Menicon Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MCOK-01
Record Dates: First submitted 2023-08-23; First posted 2023-09-14 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-02

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | Unapproved Device: Yes | US Export: No

ARMS (2):
- Treatment (Experimental): Randomized to Treatment
  Interventions: Device: Test orthokeratology lens
- Control (Active Comparator): Randomized to Control
  Interventions: Device: Control orthokeratology lens

INTERVENTIONS:
Device: Test orthokeratology lens — Randomized to test orthokeratology lens worn during sleep every night
  Arms: Treatment
Device: Control orthokeratology lens — Randomized to control orthokeratology lens worn during sleep every night
  Arms: Control

SUMMARY:
A prospective, multicenter, randomized, controlled clinical trial of orthokeratology lens

DETAILED DESCRIPTION:
The test product is the orthokeratology lens, and the control product is a commercially available orthokeratology lens. The number of enrolled subjects is 390, and clinical observation is performed for 12 months.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with myopia and myopic astigmatism
2. Those who are not willing to wear glasses in daily life
3. Fully understand of the purpose of the clinical trial and agree to sign the informed consent form to participate in clinical trials, based on his/her willingness
4. Those who can visit the institution on scheduled dates
5. Those who can receive guidance and tests as required by the investigator
6. Those who fully understand and follow the instructions of the lenses for this clinical trial

Exclusion Criteria:

<At screening>

1. Best corrected vision acuity of less than 0.8 with spectacles
2. Subjective refraction test shows spherical power greater than -6.00D，less than -0.50D or astigmatism greater than 1.5D
3. Patients in need of treatment for eye disease other than refractive error (excluding those receiving artificial tears eye drops due to the wearing of corneal contact lenses)
4. The medical history of intraocular surgery that may affect the effect of wearing the lens for this clinical trial (those with corneal transplantation, Retinal detachment, etc.)
5. The medical history of refractive corneal surgery
6. Those in need of a strength out of the scope of lens for this clinical trial
7. Having eye allergic diseases that may cause disorders in wearing the lenses for this clinical trial
8. All Corneal abnormalities including keratoconus, corneal dystrophy, previous history of ocular herpes infections, acute dry eyes, low corneal endothelial cell counts.
9. Pregnant (judgment according to her known information) or those who plan to become pregnant during clinical trial, or those who are breast feeding
10. Those who are participating in other clinical trials or have participated in other clinical trial in the past 30 days
11. Prior experience with use of rigid lenses within the previous 3 weeks or use of soft lenses within the previous 3 days
12. Prior experience with myopia control treatment (e.g. atropine, orthokeratology, multifocal soft contact lenses)
13. Minor/adult subjects who lack mental capacity
14. Other not suitable for this clinical trial at investigator's discretion <At the beginning of the wearing>

(1) Those who are determined to be unable to obtain good centralized positioning even though changing strength (2) Pregnancy confirmed (3) Those who are difficult in continuing the clinical trial at investigator's discretion

Ages: 6 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 390 (Actual)
Dates: Start 2022-07-29 (Actual); Primary Completion 2024-10-31 (Actual); Study Completion 2024-10-31 (Actual)

PRIMARY OUTCOMES:
Visual acuity | 1 year
  uncorrected visual acuity measured using logMAR chart
Axial length | 1 year
  axial eye length in millimeter measured by MYAH (Topcon) and IOL master (ZEISS)
Refraction | 1 year
  spherical and cylinder power in diopter for best corrected visual acuity measured subjectively

SECONDARY OUTCOMES:
Adverse Events | 1 year
  Adverse events are classified into moderate, middle, or severe.

CONTACTS AND LOCATIONS:
Overall Officials: Stan Isaacs, Study Director — I & Vision Research Centre Pte. Ltd.
Locations (3):
- Singapore (3):
  - I&VISION Research Centre, Singapore
  - Myopia Specialist Centre, Singapore
  - Stan Isaacs, Singapore